CLINICAL TRIAL: NCT02914366
Title: Ambroxol as a Novel Disease Modifying Treatment for Parkinson's Disease Dementia
Brief Title: Ambroxol as a Treatment for Parkinson's Disease Dementia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Weston Brain Institute (Other); Western University, Canada (Other); London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Stephen Pasternak, M.D., Ph.D., Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R15-006; 105234 (Other: Western University Health Science Research Ethics Board (HSREB)); 181033 (Other: Health Canada)
Record Dates: First submitted 2016-09-08; First posted 2016-09-26 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease Dementia
Keywords: Ambroxol; Dementia; Parkinson's disease; Disease modifying treatment; Pharmacological Chaperone; GBA1
MeSH Terms: conditions — Dementia; Parkinson Disease | interventions — Ambroxol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambroxol high dose (1050 mg) (Experimental): Participants randomized to the 1050 mg/day group will begin with a dose of 225mg (3 mg/kg/day), increasing bi-weekly by ~3mg/kg to a dose of 1050 mg/day (~l5 mg/kg/day).
  Interventions: Drug: Ambroxol
- Placebo (Placebo Comparator): Participants receive capsules visually identical to the experimental groups but without active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ambroxol
  Other Names: Mucosolvon
  Arms: Ambroxol high dose (1050 mg)
Other: Placebo
  Arms: Placebo

SUMMARY:
The present study will test the hypothesis that the medication Ambroxol is safe and well tolerated and will improve cognitive and motor symptoms of Parkinson's Disease Dementia (PDD). Ambroxol has been shown to raise the levels of the enzyme beta-glucocerebrosidase resulting in lower the levels of the protein alpha-synuclein, both of which have been shown to improve cognition in mouse models. This will be a 52 week trial of Ambroxol in 75 individuals with PDD. Participants will undergo clinical, neuropsychological and neuroimaging assessment throughout the study to assess changes.

DETAILED DESCRIPTION:
The increasing prevalence of dementia is a serious threat to the medical system and society. About 500,000 Canadians are affected with dementia, and this number will rise to more than 1 million in the next 20 years. Dementia already costs the Canadian economy 15 billion dollars per year. While much of the focus of dementia is on Alzheimer's disease, autopsy studies suggest that up to 30% of dementia is due to diseases caused by abnormal alpha-synuclein accumulation (Synucleinopathies) such as Parkinson's Disease Dementia (PDD). People with Parkinson's disease (PD) typically present with motor symptoms, but the disease is also characterized by insidious cognitive decline, increasing in relation to disease duration. Glucocerebrosidase (GCase) is a degradative enzyme that resides in a subcellular compartment called the lysosome, and cleaves a neutral glycolipid, glucocerebroside, present in the plasma membrane of most cells. GCase is intimately linked with PD. Being an "asymptomatic carrier" of a GCase mutation is currently the highest genetic risk factor for PD, with some studies suggesting up to 1/3 of patients carry mutations.

Reductions in GCase activity most likely also plays a role in sporadic PD, as these patients have lower levels of GCase in their brain and cerebrospinal fluid, even when they do not carry a mutant GCase allele. Reducing GCase genetically or pharmacologically in animal studies results in cognitive impairment. The aggregates causing the impairment can be cleared by re-introduction of normal GCase back into the brain. In addition, overexpressing GCase in the brain of a PD mouse model improves cognition. GCase therefore appears to be an excellent target for a therapy that addresses the underlying pathophysiology of PDD to improve or stop disease progression.

Ambroxol is an expectorant that has been available over the counter in more than 50 countries for over 30 years. Recently, the Mahuran Lab identified Ambroxol by screening a library of compounds as an agent that stabilizes wild-type (normal) GCase. By stabilizing GCase, Ambroxol is able to markedly increase GCase protein and activity in normal and Gaucher disease fibroblasts at doses of 10 micromolar. Ambroxol can also increase GCase in normal mouse neuronal cultures to more than 150% of normal at a dose of 30 micromolar. Ambroxol has good lipophilicity (cLogP = 2.8) and low polar surface area (PSA 58 Å2), predicting good CNS penetration. Unpublished studies performed by ExSAR corporation demonstrate that in single and multiple dose experiments in rats, Ambroxol crossed rapidly into the brain and exhibited brain to plasma concentration ratios of greater than 10 indicating outstanding CNS penetration. Ambroxol has an excellent safety record, and has been studied in >15,000 patients in more than 100 trials. Ambroxol is sold over the counter in much of the world as an expectorant at doses of 75-120 mg/day. Furthermore, Ambroxol is considered so safe that it is approved for intravenous use in pregnant women at a dose of 1000 mg/day IV (15 mg/kg) to improve fetal lung maturation before preterm delivery. Clinical trials in more than 390 pregnant women have been performed using doses up to 3000 mg in one day and 1300 mg/day for up to 33 days. Critically ill neonates have also been given doses as high as 30 mg/kg for respiratory distress. The fact that Ambroxol has been used at very high doses in pregnant women and neonates suggests that these doses are safe. In pilot studies, Ambroxol was effective at improving GCase function in humans. In a trial aimed at non-neurological Gaucher disease, 12 patients received 150 mg/day for 6 months, and all but one had some measureable improvement. The best response was in the lightest patient (who received 3 mg/kg/day), suggesting that Ambroxol was under dosed. Ambroxol has also been administered to three Japanese Gaucher disease patients with severe neurological disease, at 1000-3000 mg/day for 12-31 months. These patients had improvements in seizure frequency and neurological symptoms; one patient regained the ability to sit unsupported and to walk.

Ambroxol has never been examined in PD or Lewy Body Dementia patients; however, trials of pharmacological chaperone therapy have been suggested in a recent review in the journal "The Proceedings of the National Academy of Sciences." A successful outcome of this trial will greatly accelerate the development of therapeutics for neurodegenerative disease. This proposal outlines a completely novel pharmacological target for PDD, namely the enzyme GCase. It also proposes a completely novel therapy using the drug Ambroxol, an agent considered safe enough to give to pregnant women, which has improved GCase function in pilot studies in humans. This strategy could stop or reverse the underlying pathology of PD; it might allow patients to get better. Furthermore, re-purposing an existing medication with excellent safety record will greatly shorten the time to bring this therapy to general use, allowing us to leapfrog the normally decades-long drug development process.

This study will test the hypothesis that Ambroxol can improve the course of cognitive impairment or motor function in PDD by raising GCase levels in blood and CSF. The study specific aims will be 1) to demonstrate the efficacy of Ambroxol in improving, or slowing the progression of cognitive deficits, motor symptoms, or CSF/neuroimaging biomarkers, 2) to acquire additional pharmacokinetic and pharmacodynamic data for use in future trials and 3) to demonstrate the safety and tolerability of Ambroxol in patients with PDD.

This study is a randomized, placebo-controlled, double-blind trial of Ambroxol 1050 mg/day in individuals with mild to moderate PDD. Participants will be allowed but not required to be receiving concomitant treatment in a stable regimen for Parkinson's disease and dementia. Eligibility for enrollment will be assessed initially at one or more Screening visits, which are to occur within 28 days of Baseline. Eligible subjects will be randomly assigned (1:1) at the Baseline visit to one of the following two groups: Ambroxol 1050 mg/day or placebo.

Patients will be randomized to receive placebo or Ambroxol (1050mg). Participants randomized to Ambroxol group will begin with a dose of 225mg (3 mg/kg/day), increasing bi-weekly by ~3mg/kg to a dose of 1050 mg/day (~l5 mg/kg/day).

After 52 weeks, all patients will be offered a 6-month open label extension of Ambroxol 1050 mg/day.

For minor AE's (e.g. GI upset), patients will be allowed to spread the medication dose over a longer interval, or to reduce the dose to the highest dose tolerated. The dose can be advanced again after 2 weeks. For significant but non-threatening laboratory abnormalities, doses can be reduced to the highest dose tolerated. Patients will be allowed to stop taking medication if there is concern about a drug reaction of a clinically significant alteration in laboratory values. They can be re-challenged 2-4 weeks after these abnormalities have resolved.

If one experiences a severe allergic reaction that is possibly related to the study medication, the participant will be discontinued from the trial.

The dose-plasma level and plasma concentration-response relationships will be assessed by measuring plasma Ambroxol levels and lymphocyte GCase at baseline and 2 weeks after each dose escalation. At 12 weeks, blood and CSF Ambroxol and GCase activity will be quantitated. Patients will be followed at weeks screening, baseline, week 2, 4, 6, 8, 12, 18, 26, 34, 42 and 52 for blood work, ECG,and interview. Physical exam occurs at all visits except week 2 and 8. Neurological examinations occur at baseline, and weeks 6, 12, 18, 34, 42 and 52. Neuropsychological exam and movement testing will take place at baseline, week 26 and week 52. An MRI will be performed at screening and week 52. CSF will be collected at baseline, week 12 and week 52.

Patients will undergo clinical neuropsychological assessment at baseline, week 26, and week 52. At each assessment they will be administered standard tests of cognition such as the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog), ADCS-Clinician's Global Impression of Change (CGIC), Parkinson Disease-Cognitive Rating Scale (PD-CRS), Clinical Dementia Rating Scale (CDR), Montreal Cognitive Assessment (MoCA), Trail Making Test (TRAILS), Stroop, Geriatric Depression Scale (GDS), Neuropsychological Inventory (NPI); and tests of motor function/Parkinsonism such as the motor subscale of UPDRS and Quantitative Movement Testing, including Purdue Pegboard, Timed up and Go, and gait kinematics. MRI will be performed during screening and week 52. Mini-Mental Status Exam (MMSE) will be performed at all visits except weeks 2 and 8. A lumbar puncture will be performed at Baseline, week 12 and week 52.

The Primary Outcome measures will be the: ADAS-cog and the CGIC. These are standard cognitive and clinical measures used in almost all cognitive clinical trials. Secondary/ Exploratory outcome measures will include

1. Standard tests of cognition such as the MMSE, MoCA, CDR, , TRAILS, NPI, PD-CRS
2. Tests of motor function/Parkinsonism: UPDRS, Purdue Pegboard, Timed Up and Go, and Quantitative Movement Testing
3. CSF and Neuroimaging biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Age >50,
2. Mild to Moderate Dementia (established by an upper cut off of a Montreal Cognitive Assessment score of 24 or below, and the lower bound by a Mini Mental State Exam of 16 or greater),
3. Parkinson's Disease (Hoehn & Yahr stage 2 - 3.5) clearly established more than 1 year before the onset of dementia
4. Patients must have a responsible caregiver = 4 days/wk
5. Must be on stable doses of medications for Parkinson's disease mood and cognition (Cholinesterase Inhibitor) for at least 3 months prior to the study.

Exclusion Criteria:

1. Evidence of clinically significant stroke or other neurological condition
2. Any other serious underlying condition (i.e. cancer or unstable cardiac disease etc.
3. Concurrent treatment with oral anticoagulants (including Vitamin K agonists and Novel Oral Anticoagulants (NOACs)) within 4 weeks of screening or anticipated during the 52 week double-blind and open label periods. Specifically, Apixaban, Dabigatran, Edoxaban, Fondaparinux, Rivaroxaban, and Warfarin are prohibited concomitant medications.

3.1 Exceptions: antiplatelet agents such as Aspirin, Clopidogrel, and Aggrenox are allowed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) | baseline, week 26, and week 52
  This 70-point test examines language, recall, word finding, comprehension, naming, drawing, praxis, orientation, and word recognition. Although designed for Alzheimer's disease where it is considered a gold standard, the ADAS-Cog has been used effectively in many clinical trials of PDD including large randomized trials. This scale has been recommended for the assessment of Parkinson's dementia in "Diagnostic Procedures for Parkinson's Disease Dementia: Recommendations from the Movement Disorder Society Task Force"
Changes in the ADCS-Clinician's Global Impression of Change (CGIC) | baseline, week 26, and week 52
  This is a 7-point scale for rating patient function in cognition behavior and activities of daily living, and this test is standard in clinical trials in Alzheimer's disease and has been useful in trials with PDD.

SECONDARY OUTCOMES:
Changes in the Montreal Cognitive Assessment | baseline, week 26, and week 52
Changes in the Clinical Dementia Rating Scale (CDR) | baseline, week 26, and week 52
Changes in the Trail Making Test (TRAILS) | baseline, week 26, and week 52
Changes in the Parkinson's Disease-Cognitive Rating Scale (PD-CRS) | baseline, week 26, and week 52
Changes in the Stroop Test | baseline, week 26, and week 52
Changes in the Unified Parkinson's disease Rating Scale motor subsection (UPDRS-III) | baseline, week 26, and week 52
Changes in the Purdue Pegboard | baseline, week 26, and week 52
Changes in the Timed Up and Go | baseline, week 26, and week 52
Change in Quantitative Movement Testing | baseline, week 26, and week 52
  gait assessment on electronic mat (Zeno Walkway System)
Changes in Cerebrospinal Fluid (CSF) biomarkers | baseline, week 12, and week 52
  levels of α-synuclein (pg/ml), Tau (pg/ml), phospho-Tau (pg/ml) and beta amyloid-42 (pg/ml)
Changes in Magnetic Resonance Imaging (MRI) | baseline and week 52
  brain ventricle volume (cm3) and hippocampal atrophy (cm3)
Changes in the Mini-Mental State Examination | screening, baseline, week 4, week 6, week 12, week 18, week 26, week 34, week 42, week 52
Changes in GCAse in lymphocytes | baseline, week 2, week 4, week 6, week 8, week 12, week 18, week 26, week 34, week 42, week 52
  from blood sample
Changes in Plasma Ambroxol levels | baseline, week 2, week 4, week 6, week 8, week 12, week 18, week 26, week 34, week 42, week 52
  from blood sample
Mayo Fluctuation Questionnaire | baseline, week 26, and week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Peer reviewed publication | Presentation

REFERENCES:
- [Background] Lang AE, Obeso JA. Challenges in Parkinson's disease: restoration of the nigrostriatal dopamine system is not enough. Lancet Neurol. 2004 May;3(5):309-16. doi: 10.1016/S1474-4422(04)00740-9. PMID 15099546
- [Background] Balducci C, Pierguidi L, Persichetti E, Parnetti L, Sbaragli M, Tassi C, Orlacchio A, Calabresi P, Beccari T, Rossi A. Lysosomal hydrolases in cerebrospinal fluid from subjects with Parkinson's disease. Mov Disord. 2007 Jul 30;22(10):1481-1484. doi: 10.1002/mds.21399. PMID 17546678
- [Background] Gegg ME, Burke D, Heales SJ, Cooper JM, Hardy J, Wood NW, Schapira AH. Glucocerebrosidase deficiency in substantia nigra of parkinson disease brains. Ann Neurol. 2012 Sep;72(3):455-63. doi: 10.1002/ana.23614. PMID 23034917
- [Background] Sardi SP, Clarke J, Viel C, Chan M, Tamsett TJ, Treleaven CM, Bu J, Sweet L, Passini MA, Dodge JC, Yu WH, Sidman RL, Cheng SH, Shihabuddin LS. Augmenting CNS glucocerebrosidase activity as a therapeutic strategy for parkinsonism and other Gaucher-related synucleinopathies. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3537-42. doi: 10.1073/pnas.1220464110. Epub 2013 Jan 7. PMID 23297226
- [Background] Malerba M, Ragnoli B. Ambroxol in the 21st century: pharmacological and clinical update. Expert Opin Drug Metab Toxicol. 2008 Aug;4(8):1119-29. doi: 10.1517/17425255.4.8.1119. PMID 18680446
- [Background] Maegawa GH, Tropak MB, Buttner JD, Rigat BA, Fuller M, Pandit D, Tang L, Kornhaber GJ, Hamuro Y, Clarke JT, Mahuran DJ. Identification and characterization of ambroxol as an enzyme enhancement agent for Gaucher disease. J Biol Chem. 2009 Aug 28;284(35):23502-16. doi: 10.1074/jbc.M109.012393. Epub 2009 Jul 3. PMID 19578116
- [Background] Luan Z, Li L, Higaki K, Nanba E, Suzuki Y, Ohno K. The chaperone activity and toxicity of ambroxol on Gaucher cells and normal mice. Brain Dev. 2013 Apr;35(4):317-22. doi: 10.1016/j.braindev.2012.05.008. Epub 2012 Jun 7. PMID 22682976
- [Background] Laoag-Fernandez JB, Fernandez AM, Maruo T. Antenatal use of ambroxol for the prevention of infant respiratory distress syndrome. J Obstet Gynaecol Res. 2000 Aug;26(4):307-12. doi: 10.1111/j.1447-0756.2000.tb01327.x. PMID 11049243
- [Background] Luerti M, Lazzarin A, Corbella E, Zavattini G. An alternative to steroids for prevention of respiratory distress syndrome (RDS): multicenter controlled study to compare ambroxol and betamethasone. J Perinat Med. 1987;15(3):227-38. doi: 10.1515/jpme.1987.15.3.227. PMID 3323457
- [Background] Wauer RR, Schmalisch G, Hammer H, Buttenberg S, Weigel H, Huth M. Ambroxol for prevention and treatment of hyaline membrane disease. Eur Respir J Suppl. 1989 Mar;3:57S-65S. PMID 2662997
- [Background] Schmalisch G, Wauer RR, Bohme B. Changes in pulmonary function in preterm infants recovering from RDS following early treatment with ambroxol: results of a randomized trial. Pediatr Pulmonol. 1999 Feb;27(2):104-12. doi: 10.1002/(sici)1099-0496(199902)27:23.0.co;2-t. PMID 10088933
- [Background] Narita A, Kubota N, Takayama R, Takahashi Y, Maegaki Y, Suzuki Y, & Ohno K. Chaperone therapy for neuronopathic Gaucher disease. Molecular Genetics and Metabolism, 108(2): S69, 2013.
- [Background] Abstracts of the 12th International Child Neurology Congress and the 11th Asian and Oceanian Congress of Child Neurology. May 27-June 1, 2012. Brisbane, Australia. Dev Med Child Neurol. 2012 Jun;54 Suppl 4:5-220. No abstract available. PMID 22606700
- [Background] Zimran A, Altarescu G, Elstein D. Pilot study using ambroxol as a pharmacological chaperone in type 1 Gaucher disease. Blood Cells Mol Dis. 2013 Feb;50(2):134-7. doi: 10.1016/j.bcmd.2012.09.006. Epub 2012 Oct 22. PMID 23085429
- [Derived] Silveira CRA, Coleman KKL, Borron K, Tirona RG, Rupar CA, Zou G, Hegele RA, Wellington C, Stukas S, Finger EC, Bartha R, Morrow SA, Wells JL, Borrie MJ, Mahuran D, MacDonald PA, Jenkins ME, Jog MS, Dresser G, Fox S, Camicioli R, Feagan B, Mendonca DA, Mayich M, Sharma MD, Pandey SK, Pasternak SH. Ambroxol as a Treatment for Parkinson Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2025 Jun 30;82(8):797-807. doi: 10.1001/jamaneurol.2025.1687. Online ahead of print. PMID 40587145
- [Derived] Silveira CRA, MacKinley J, Coleman K, Li Z, Finger E, Bartha R, Morrow SA, Wells J, Borrie M, Tirona RG, Rupar CA, Zou G, Hegele RA, Mahuran D, MacDonald P, Jenkins ME, Jog M, Pasternak SH. Ambroxol as a novel disease-modifying treatment for Parkinson's disease dementia: protocol for a single-centre, randomized, double-blind, placebo-controlled trial. BMC Neurol. 2019 Feb 9;19(1):20. doi: 10.1186/s12883-019-1252-3. PMID 30738426